CLINICAL TRIAL: NCT03058653
Title: Use of a Mini-fluid Bolus to Identify Fluid Responsiveness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017CRI89
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Output, Low; Cardiac Output, High
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients (Experimental): Small fluid boluses - The first 250ml of fluid will be given in 50ml boluses using a 50ml syringe
  Interventions: Procedure: Small fluid boluses of 50 ml; Device: LIDCORapid Monitor

INTERVENTIONS:
Procedure: Small fluid boluses of 50 ml — Participants will receive small 50ml boluses of fluid up to 250ml in total. The remainder will be given as infusion pump method at a rate of 1000ml/hour which will complete in 15 minutes. In total, the 500ml will be given over 25 minutes.
Device: LIDCORapid Monitor — Addition of the LIDCORapid Monitor to measure stroke volume

SUMMARY:
On the Intensive Care Unit doctors give a lot of fluid to patients in order to improve their blood pressure, amount of urine made or to let doctors stop drugs that are needed to keep blood pressure up. Doctors normally give patients 500ml of fluid over 25 minutes as standard, however it is very difficult to know if giving those fluids and how much fluid will help (it does in some but not others). If a person gets too much fluid this can also cause problems such as fluid in lungs, poor kidney function, or swelling in the limbs.

The LidCo Rapid monitor lets the Intensive Care Unit (ICU) team know the amount of blood the heart pushes out with each beat (Stroke volume). It works by following the tracing off the arterial line (Blood pressure monitor) that has been inserted as part of the standard care of a patient on the ICU. It does not need any other invasive procedures or drug administration to work.

This study is using this monitor to see if it can identify a method of improving the administration of intravenous fluids on the Intensive Care Unit. The study is looking to see if it can identify whether giving a small amount of fluid first identifies people who will benefit from more fluid and those that won't.

DETAILED DESCRIPTION:
Adult patients whom the Consultant Intensivist decides should receive a fluid challenge as part of their standard care in order to improve haemodynamic parameters will be approached. Reasons for fluid administration include evidence of inadequate tissue perfusion such as raised blood lactate or poor urine output, hypotension or attempts to wean vasopressor dose.

Patients will be identified as suitable for inclusion by the Consultant Responsible for the Intensive Care Unit on each day. As fluid responsiveness is a transient phenomenon which disappears after significant fluid resuscitation it is proposed that patients will be immediately entered into the study so that the study contains a mix of fluid responsive and non-responsive patients in order to get the time critical data required which may be lost if there is a significant delay before study entry. Informed consent will be sought from the patient, or if they are incapacitated by critical illness, their relative will be approached for assent as soon as possible and within 48 hours of study enrollment. This is in line with recommendations for Research involving emergency treatment.

The LiDCOrapid machine will be connected in the same manner as the LiDCOplus machine, currently in use on ICU, in order to obtain the stroke volume measurement. A smartcard is inserted and the patient details entered. Monitoring will continue until fluids are clinically indicated. Patients will be given fluid boluses via either peripheral or central venous catheters.

The following data will be collected for each patient:

Age, Gender, Height, Weight, diagnosis requiring ICU admission, location of venous and arterial catheters, APACHE II scores, Cumulative fluid balance at time of bolus administration, Ventilation status (self-ventilating, non-invasive ventilation, invasive ventilation and mode if appropriate), tidal volume if measured, drugs being infused (sedatives, inotropes, vasoactive drugs, diuretics, muscle relaxants, etc), presence of renal replacement therapy.

Fluid administration protocol:

Patients will be monitored just prior to infusion for hemodynamic stability, Standard practice is to administer a bolus of 500ml given via an infusion pump at a rate of 1200mL/hour (25min).

For study patients the first 250ml will be given in 50ml boluses using a 50ml syringe. Each bolus will be given over approximately 1 minute and the study measurements will be recorded followed by a wait for response of 1 minute. This will be repeated for each subsequent bolus until 250ml has been given (i.e. 5 boluses). The remaining 250ml will be given via the standard infusion pump method at a rate of 1000ml/hour which will complete in 15 minutes. In total, the 500ml will be given over 25 minutes.

At the end of each bolus Stroke volume, cardiac output, heart rate, blood pressure will be determined.

Up to 2 sets of data per patient per day will be collected. The majority of patients routinely stay in the ICU for 2 days, while in a smaller group, for much longer. A maximum of 4 data sets will be collected per patient. The fluid boluses will be administered at the discretion of the treating physician who believes that they will improve the clinical condition of the patient. The study team will have no influence on the timing of these.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients whom the Consultant Intensivist decides should receive a fluid challenge as part of their standard care in order to improve haemodynamic parameters

Exclusion Criteria:

* Age under 18
* severe haemodynamic instability
* persistent arrhythmia (including atrial fibrillation)
* pregnant patients
* palliative care only patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
stroke volume | 1 minute intervals for 10 mins, then at 25 mins over 4 episodes in 2 days
  measurement of stroke volume after each bolus of fluid has been given
Cardiac out-put | 1 minute intervals for 10 mins, then at 25 mins over 4 episodes in 2 days
  If Cardiac output increased by 15% then the patient is defined as a "fluid responder" and should receive more fluid. If there is not a 15% increase, then the patient will have no benefit from further fluid loading.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew MacDuff, Principal Investigator — The Royal Wolverhampton NHS Trust

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available